CLINICAL TRIAL: NCT01298089
Title: LASIK Flap Thickness Predictability With the Carriazo Pendular Microkeratome
Brief Title: A Study of Flap Thickness Results Using the Carriazo Pendular Microkeratome - 130 Micrometers Head.
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Eleftherios Paschalis / PhD, Eye Institute of Thrace / Democritus University
Other Study IDs: Carriazo Pendular
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Corneal Flap Thickness (Micrometers)
Keywords: Flap; LASIK; Corneal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Device: Carriazo Pendular microkeratome

SUMMARY:
A study of flap thickness predictability in patients submitted to Laser in Situ Keratomileusis (LASIK) with the Carriazo-Pendular microkeratome (130 micrometers head size).

ELIGIBILITY:
Inclusion Criteria:

* LASIK candidates treated with the Carriazo-Pendular microkeratome - 130 micron head

Exclusion Criteria:

* corneal irregularities > 3D
* Thin corneal CCT < 460μm
* Active anterior segment disease
* Previous intraocular or corneal surgery
* History of herpetic eye disease
* Corneal scarring
* Glaucoma
* Severe dry eye
* Topographic evidence of keratoconus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients submitted to LASER refractive correction at the Eye Institute of Thrace, Democritus University
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Corneal flap thickness (micrometers) | 6 months postoperatively
  Flap thickness was calculated by subtracting the preoperative central corneal thickness minus the intraoperative residual stromal thickness. All measurements were made using ultrasound pachymetry (non-interventional technique).

CONTACTS AND LOCATIONS:
Locations (1):
- Eleftherios Paschalis, Alexandroupoli, Euros, Greece

REFERENCES:
- [Background] Paschalis EI, Aristeidou AP, Foudoulakis NC, Razis LA. Corneal flap assessment with Rondo microkeratome in laser in situ keratomileusis. Graefes Arch Clin Exp Ophthalmol. 2011 Feb;249(2):289-95. doi: 10.1007/s00417-010-1433-7. Epub 2010 Jun 25. PMID 20577755
- [Background] Alio JL, Pinero DP. Very high-frequency digital ultrasound measurement of the LASIK flap thickness profile using the IntraLase femtosecond laser and M2 and Carriazo-Pendular microkeratomes. J Refract Surg. 2008 Jan;24(1):12-23. doi: 10.3928/1081597X-20080101-03. PMID 18269144
- [Background] Kymionis GD, Portaliou DM, Tsiklis NS, Panagopoulou SI, Pallikaris IG. Thin LASIK flap creation using the SCHWIND Carriazo-Pendular microkeratome. J Refract Surg. 2009 Jan;25(1):33-6. doi: 10.3928/1081597X-20090101-06. PMID 19244951